CLINICAL TRIAL: NCT01441401
Title: Special Investigation Of Gabapen For Pediatric (Regulatory Post Marketing Commitment Plan)
Brief Title: Safety and Efficacy of Gabapen for Pediatric (Regulatory Post Marketing Commitment Plan)
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A9451175
Record Dates: First submitted 2011-09-23; First posted 2011-09-27 (Estimated); Results first posted 2016-10-06 (Estimated); Last update posted 2021-02-03 (Actual); Status verified 2016-08

CONDITIONS: Epilepsies, Partial
Keywords: Gabapentin; Epilepsies; safety
MeSH Terms: conditions — Epilepsies, Partial; Epilepsy | interventions — Gabapentin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Gabapentin: Peadiatric subjects taking Gabapen Tablets and syrup.
  Interventions: Drug: gabapentin

INTERVENTIONS:
Drug: gabapentin — According to Japanese Package Insert: For infants and children aged 3 to 12 years, a daily dosage of 10 mg/kg of gabapentin should be administered orally in 3 divided doses on the first day of treatment, and an effective dosage of 20 mg/kg should be administered to them in 3 divided doses on day 2. From day 3 on, infants aged 3 to 4 years should be maintained on the dosage of 40 mg/kg, and children aged 5 to 12 years on the dosage of 25 to 35 mg/kg administered orally in 3 divided doses, respectively (the maximum daily dosage: 1800 mg). Though the maintenance dosage may be adjusted depending on the patient's condition, the maximum daily dosage should be 50 mg/kg. At any time point, dosage should not exceed that the dosage for adults and children aged 13 years.As for children aged 13 years or over is as same as administration for adult.

SUMMARY:
This investigation aims to understand the following issues in pediatric patients, as well as to assess the need of a special investigation and a post-marketing clinical study:

* The frequency of treatment related adverse events.
* The frequency of efficacy assessment.
* Treatment related unlisted adverse events in Japanese Package Insert.
* Risk factors likely to affect the frequency of treatment related adverse event.

DETAILED DESCRIPTION:
All the patients whom an investigator prescribes the first gabapentin should be registered consecutively until the number of subjects reaches target number in order to extract patients enrolled into the investigation at random.

ELIGIBILITY:
Inclusion Criteria:

* All the pediatric subjects (aged 3-15 years) whom an investigator prescribes the first gabapentin (tablets, syrup, and switch to syrup from tablet) should be registered consecutively until the number of subjects reaches target number in order to extract patients enrolled into the investigation at random.

Exclusion Criteria:

* Patients who have been enrolled in the drug use investigation of Gabapen tablets in adults (protocol No. A9451163).
* Patients who receive Gabapen tablets or syrup before, except for switched from tablets to syrup.

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study whom an investigator involving A9451175 prescribes the Gabapentin
Sampling Method: Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2011-12; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9451175&StudyName=Safety%20and%20Efficacy%20of%20Gabapen%20for%20Pediatric%20%28Regulatory%20Post%20Marketing%20Commitment%20Plan%29

RESULTS

PARTICIPANT FLOW:
Groups:
- Gabapentin Tablets/Syrup: For participants aged 13 years or older, 600 mg in 3 divided doses (div.) was administered on day 1 and an effective dose of 1200 mg in 3 div. was administered on day 2. From day 3 on, participants were maintained on 1200 mg to 1800 mg in 3 div. The maintenance dose was adjusted according to the symptoms (up to a maximum daily dose of 2400 mg). For participants aged 3 to 12 years, 10 mg/kg/day was administered orally in 3 div. on day 1 of the treatment, and an effective dose of 20 mg/kg/day was administered in 3 div. on day 2. From day 3 on, participants aged 3 to 4 years were maintained on 40 mg/kg/day in 3 div. and participants aged 5 to 12 years were maintained on 25 to 35 mg/kg/day in 3 div. The maintenance dose was adjusted according to the symptoms (up to a maximum dose of 50 mg/kg/day). At any time point, the dose was not exceeded that for participants aged 13 years or older.
Period: Overall Study
Arm/Group | Gabapentin Tablets/Syrup
Started | 82
Completed | 82 (Number of participants whose survey form was collected was presented.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Gabapentin Tablets/Syrup
Number analyzed (Participants) | 82
Age, Customized [Number; unit: Participants] — Participants taking gabapentin tablets/syrup according to the Japanese package insert.
  Participants
    3 to 4 years | 14
    5 to 12 years | 54
    13 to 15 years | 14
Sex: Female, Male [Count of Participants; unit: Participants] — Participants taking gabapentin tablets/syrup according to the Japanese package insert.
  Participants
    Female | 39
    Male | 43

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Related Adverse Events
Description: A treatment-related adverse event was any untoward medical occurrence attributed to gabapentin in a participant who received gabapentin. Relatedness to gabapentin was assessed by the investigator and sponsor (Pfizer Japan Inc.).
Time Frame: MAX 104 weeks
Population: The safety analysis population comprised of participants who had met the inclusion criteria and had taken gabapentin at least once.
Measure: Number; unit: Participants
Arm/Group | Gabapentin Tablets/Syrup
Number analyzed (Participants) | 82
Participants | 5

2. Primary Outcome: Clinical Efficacy Rate
Description: Clinical efficacy rate, which was defined as the percentage of participants who achieved clinical efficacy over the total number of efficacy analysis population, was presented along with the corresponding exact 2-sided 95% CI. For the basis of efficacy evaluation, frequencies of epileptic seizure were recorded during the previous 4 weeks from the treatment start date, and that from the end date of assessment period. Clinical efficacy was assessed according to the following categories: (1) effective, (2) not effective, or (3) not assessable.
Time Frame: MAX 104 weeks
Population: The analysis population comprised of the participants in the efficacy analysis population from which those with data not assessable were excluded. n=number of participants with assessable data at each post-baseline time point.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Gabapentin Tablets/Syrup
Number analyzed (Participants) | 75
Percentage of participants
  Week 12 (n = 73) | 56.2 [44.1 to 67.8]
  Week 52 (n = 52) | 57.7 [43.2 to 71.3]
  Week 104 (n = 14) | 64.3 [35.1 to 87.2]
  End of assessment period (n = 66) | 42.4 [30.3 to 55.2]

3. Secondary Outcome: Number of Participants With Treatment-Related Adverse Events Unexpected From Japanese Package Insert
Description: A treatment-related adverse event was any untoward medical occurrence attributed to gabapentin in a participant who received gabapentin. Expectedness of the adverse event was determined according to the Japanese package insert. Relatedness to gabapentin was assessed by the investigator and sponsor (Pfizer Japan Inc.).
Time Frame: MAX 104 weeks
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Gabapentin Tablets/Syrup
Number analyzed (Participants) | 82
Participants | 0

4. Secondary Outcome: Number of Participants With Risk Factors for Treatment-Related Adverse Events
Description: A treatment-related adverse event was any untoward medical occurrence attributed to gabapentin in a participant who received gabapentin. Participants with treatment-related adverse events were counted by each candidate risk factor (including gender, age, and disease eligible for the survey) to assess whether these were risk factors for the treatment-related adverse events. No inferential analyses of risk factors were performed because of a small number of the events (5 events).
Time Frame: MAX 104 weeks
Population: The safety analysis population comprised of participants who had met the inclusion criteria and had taken gabapentin at least once. No data displayed because outcome measure has zero total participants analyzed.
Arm/Group | Gabapentin Tablets/Syrup
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of Participants Who Responded to Treatment With Gabapentin by Baseline Severity of Epileptic Seizure
Description: Participants who responded to the treatment with gabapentin were counted by the baseline severity of epileptic seizure (mild, moderate and severe) to assess whether the baseline severity of epileptic seizure was a factor affecting the treatment efficacy.
Time Frame: MAX 104 weeks
Population: The efficacy analysis population comprised of the participants who had at least one post-baseline efficacy evaluation for the clinical efficacy and seizure frequency in the safety analysis population. Participants with diseases not eligible for the survey were excluded from the efficacy analysis population.
Measure: Number; unit: Participants
Groups:
- Mild: Participants with mild epileptic seizure at baseline
- Moderate: Participants with moderate epileptic seizure at baseline
- Severe: Participants with severe epileptic seizure at baseline
- Unknown: Participants with unknown severity of baseline epileptic seizure
Arm/Group | Mild | Moderate | Severe | Unknown
Number analyzed (Participants) | 9 | 31 | 25 | 1
Participants | 6 | 15 | 6 | 1
Statistical Analysis 1: Comparison: Mild vs Moderate vs Severe; The factor tested was "baseline severity of epileptic seizure". The null hypothesis was that there was no association between the baseline severity of epileptic seizure (mild, moderate, and severe) and the number of participants who responded to the treatment with gabapentin; Test type: Superiority or Other; p = 0.045, Fisher Exact
Statistical Analysis 2: Comparison: Mild vs Moderate vs Severe; The factor tested was "baseline severity of epileptic seizure". The null hypothesis was that there was no ordinal trend in the number of responders to the treatment with gabapentin across the baseline severity of epileptic seizure (mild, moderate, and severe); Test type: Superiority or Other; p = 0.017, Cochran-Armitage (EXACT)

6. Secondary Outcome: Number of Participants Who Responded to Treatment With Gabapentin by Baseline Frequency of Epileptic Seizure
Description: Participants who responded to the treatment with gabapentin were counted by the baseline frequency of epileptic seizure (<=8 versus >8 episodes/per 4 weeks) to assess whether the baseline frequency of epileptic seizure was a factor affecting the treatment efficacy.
Time Frame: MAX 104 weeks
Population: as for outcome 5
Measure: Number; unit: Participants
Groups:
- <=8 Episodes: Participants with baseline episodes of epileptic seizure 8 or less
- >8 Episodes: Participants with baseline episodes of epileptic seizure more than 8
- Unknown: Participants with unknown frequency of baseline epileptic seizure
Arm/Group | <=8 Episodes | >8 Episodes | Unknown
Number analyzed (Participants) | 25 | 39 | 2
Participants | 15 | 11 | 2
Statistical Analysis 1: Comparison: <=8 Episodes vs >8 Episodes; The factor tested was "baseline frequency of epileptic seizure". The null hypothesis was that there was no difference between the baseline frequency of epileptic seizure and the number of participants who responded to the treatment with gabapentin; Test type: Superiority or Other; p = 0.018, Fisher Exact

7. Secondary Outcome: Number of Participants Who Responded to Treatment With Gabapentin by Number of Concomitant Antiepileptic Drugs at Baseline
Description: Participants who responded to the treatment with gabapentin were counted by the number of concomitant epileptic drugs at baseline across 5 categories (no drug, 1 drug, 2 drugs, 3 drugs, and 4 or more drugs) to assess whether the number of concomitant epileptic drugs at baseline was a factor affecting the treatment efficacy.
Time Frame: MAX 104 weeks
Population: as for outcome 5
Measure: Number; unit: Participants
Groups:
- No Concomitant Antiepileptic Drug: Participants taking no concomitant antiepileptic drug at baseline
- One Concomitant Antiepileptic Drug: Participants taking one concomitant antiepileptic drug at baseline
- Two Concomitant Antiepileptic Drugs: Participants taking two concomitant antiepileptic drugs at baseline
- Three Concomitant Antiepileptic Drugs: Participants taking three concomitant antiepileptic drugs at baseline
- Four or More Concomitant Antiepileptic Drugs: Participants taking four or more concomitant antiepileptic drugs at baseline
Arm/Group | No Concomitant Antiepileptic Drug | One Concomitant Antiepileptic Drug | Two Concomitant Antiepileptic Drugs | Three Concomitant Antiepileptic Drugs | Four or More Concomitant Antiepileptic Drugs
Number analyzed (Participants) | 1 | 19 | 19 | 15 | 12
Participants | 1 | 13 | 7 | 4 | 3
Statistical Analysis 1: Comparison: No Concomitant Antiepileptic Drug vs One Concomitant Antiepileptic Drug vs Two Concomitant Antiepileptic Drugs vs Three Concomitant Antiepileptic Drugs vs Four or More Concomitant Antiepileptic Drugs; The factor tested was "number of concomitant antiepileptic drugs at baseline". The null hypothesis was that there was no association between the number of concomitant antiepileptic drugs at baseline and the number of participants who responded to the treatment with gabapentin; Test type: Superiority or Other; p = 0.034, Fisher Exact
Statistical Analysis 2: Comparison: No Concomitant Antiepileptic Drug vs One Concomitant Antiepileptic Drug vs Two Concomitant Antiepileptic Drugs vs Three Concomitant Antiepileptic Drugs vs Four or More Concomitant Antiepileptic Drugs; The factor tested was "number of concomitant antiepileptic drugs at baseline". The null hypothesis was that there was no ordinal trend in the number of responders to the treatment with gabapentin across the increasing number of concomitant antiepileptic drugs at baseline; Test type: Superiority or Other; p = 0.005, Cochran-Armitage (EXACT)

8. Secondary Outcome: Number of Participants Who Responded to Treatment With Gabapentin by Treatment Period
Description: Participants who responded to the treatment with gabapentin were counted by the treatment period (non-long term [less than 1 year] or long term [1 year or more]) to assess whether the treatment period with gabapentin was a factor affecting the treatment efficacy.
Time Frame: MAX 104 weeks
Population: as for outcome 5
Measure: Number; unit: Participants
Groups:
- Non-Long Term: Participants who received gabapentin for less than 1 year
- Long Term: Participants who received gabapentin for 1 year or more
Arm/Group | Non-Long Term | Long Term
Number analyzed (Participants) | 19 | 47
Participants | 2 | 26
Statistical Analysis 1: Comparison: Non-Long Term vs Long Term; The factor tested was "treatment period with gabapentin". The null hypothesis was that there was no association between the treatment period with gabapentin and the number of participants who responded to the treatment with gabapentin; Test type: Superiority or Other; p < 0.001, Fisher Exact

9. Other Pre Specified Outcome: Number of Participants With Key Treatment-Related Adverse Events (Central Nervous System Depressant Actions)
Description: Central nervous system depressant actions including somnolence and ataxia were determined as key survey items by the sponsor (Pfizer Japan Inc.). These events were defined according to MedDRA/J version 17.1 as the events classified in "psychiatric disorders" or "nervous system disorders" of the system organ classes, or those classified in "asthenia" or "gait disturbance" of the preferred terms. A treatment-related adverse event was any untoward medical occurrence attributed to gabapentin in a participant who received gabapentin. Relatedness to gabapentin was assessed by the investigator and sponsor.
Time Frame: MAX 104 weeks
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Gabapentin Tablets/Syrup
Number analyzed (Participants) | 82
Participants | 1

10. Other Pre Specified Outcome: Number of Participants With Key Treatment-Related Adverse Events (Aggressive Behaviors)
Description: Aggressive behaviors including affect lability and hostility were determined as key survey items by the sponsor (Pfizer Japan Inc.). These events were defined as the 101 preferred terms listed by pharmaceuticals and medical devices agency and classified according to MedDRA/J version 17.1. A treatment-related adverse event was any untoward medical occurrence attributed to gabapentin in a participant who received gabapentin. Relatedness to gabapentin was assessed by the investigator and sponsor.
Time Frame: MAX 104 weeks
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Gabapentin Tablets/Syrup
Number analyzed (Participants) | 82
Participants | 1

11. Other Pre Specified Outcome: Response Ratio (R Ratio)
Description: R Ratio was calculated by the following formula, where B represented the baseline frequency of epileptic seizures during the previous 4 weeks from the treatment start date, whereas T represented the frequency of epileptic seizures during the previous 4 weeks from the end of assessment period: R Ratio = (T - B) / (T + B). R Ratio is within the range of -1 to +1, and a negative value represents a reduction in the frequency of seizure.
Time Frame: MAX 104 weeks
Population: The analysis population comprised of the participants in the efficacy analysis population who had assessable data of the frequency of epileptic seizures at the start of gabapentin treatment and at the end of assessment period. n=number of participants with assessable data at each post-baseline time point.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Gabapentin Tablets/Syrup
Number analyzed (Participants) | 73
Ratio
  Week 12 (n = 72) | -0.332 (0.458) [44.1 to 67.8]
  Week 52 (n = 56) | -0.409 (0.491) [43.2 to 71.3]
  Week 104 (n = 16) | -0.456 (0.507) [35.1 to 87.2]
  End of assessment period (n = 73) | -0.369 (0.509) [30.3 to 55.2]

12. Other Pre Specified Outcome: Responder Rate
Description: Responder rate, which was defined as the percentage of participants whose R ratio was - 0.333 or less, was presented along with the corresponding exact 2-sided 95% CI. R ratio of - 0.333 or less corresponded to the decrease of epileptic seizure frequency by 50% or more.
Time Frame: MAX 104 weeks
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Gabapentin Tablets/Syrup
Number analyzed (Participants) | 73
Percentage of participants
  Week 12 (n = 72) | 43.1 [31.4 to 55.3]
  Week 52 (n = 56) | 50.0 [36.3 to 63.7]
  Week 104 (n = 16) | 62.5 [35.4 to 84.8]
  End of assessment period (n = 73) | 49.3 [37.4 to 61.3]

13. Other Pre Specified Outcome: Reduction From Baseline in Epileptic Seizure Frequency
Description: Reduction from baseline in epileptic seizure frequency was defined by the following formula, where B represented the baseline frequency of epileptic seizures during the previous 4 weeks from the treatment start date, whereas T represented the frequency of epileptic seizures during the previous 4 weeks from the end of assessment period: Reduction from baseline in epileptic seizure frequency (%) = [(T-B) / B] X 100. The median percentages were presented along with the corresponding minimum and maximum percentages.
Time Frame: MAX 104 weeks
Population: as for outcome 11
Measure: Median (Full Range); unit: Percentage
Arm/Group | Gabapentin Tablets/Syrup
Number analyzed (Participants) | 73
Percentage
  Week 12 (n = 72) | -25.0 [-100.0 to 900.0]
  Week 52 (n = 56) | -49.0 [-100.0 to 833.3]
  Week 104 (n = 16) | -60.0 [-100.0 to 1090.5]
  End of assessment period (n = 73) | -47.9 [-100.0 to 1090.5]

ADVERSE EVENTS:
Description: The frequency of adverse events. The same event may appear as both an adverse event and a serious adverse event. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Gabapentin Tablets/Syrup
Serious Adverse Events (participants affected / at risk) | 4/82
Other Adverse Events (participants affected / at risk) | 25/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gabapentin Tablets/Syrup (N=82)
Bronchitis (Infections and infestations) | 2 (2)
Febrile convulsion (Nervous system disorders) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gabapentin Tablets/Syrup (N=82)
Influenza (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 3 (3)
Pharyngitis (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 4 (4)
Herpes zoster (Infections and infestations) | 1 (1)
Paronychia (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 12 (12)
Rhinitis (Infections and infestations) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1)
Hyperamylasaemia (Metabolism and nutrition disorders) | 1 (1)
Dissociative disorder (Psychiatric disorders) | 1 (1)
Affect lability (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Aphthous stomatitis (Gastrointestinal disorders) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.